CLINICAL TRIAL: NCT06428227
Title: A Comparison of Exercise Capacity, Respiratory Functions, and Quality of Life in Heart Failure Patients With and Without Inspiratory Muscle Weakness and Healthy Controls
Brief Title: Exercise Capacity and Fatigue in Heart Failure Patients With and Without Inspiratory Muscle Weakness
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Professor, Gazi University
Other Study IDs: GaziU5
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure
Keywords: heart failure; exercise capacity; respiratory muscle
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart failure patients with inspiratory muscle weakness: Exercise capacity (6 minute walking test), pulmonary function (spirometry), respiratory muscle strength (mouth pressure device), peripheral muscle strength (hand-held dynometer), dyspnea (The Modified Medical Research Council (MMRC) dyspnea scale), fatigue (Fatigue Severity Scale), quality of life (The Short Form 36 (SF-36) questionnaire), physical activity level (The International Physical Activity Questionnaire) were evaluated.
- Heart failure patients without inspiratory muscle weakness: Exercise capacity (6 minute walking test), pulmonary function (spirometry), respiratory muscle strength (mouth pressure device), peripheral muscle strength (hand-held dynometer), dyspnea (The Modified Medical Research Council (MMRC) dyspnea scale), fatigue (Fatigue Severity Scale), quality of life (The Short Form 36 (SF-36) questionnaire), physical activity level (The International Physical Activity Questionnaire) were evaluated.
- Healthy controls: Exercise capacity (6 minute walking test), pulmonary function (spirometry), respiratory muscle strength (mouth pressure device), peripheral muscle strength (hand-held dynometer), dyspnea (The Modified Medical Research Council (MMRC) dyspnea scale), fatigue (Fatigue Severity Scale), quality of life (The Short Form 36 (SF-36) questionnaire), physical activity level (The International Physical Activity Questionnaire) were evaluated.

SUMMARY:
In patients with heart failure, diaphragm dysfunction contributes to decreased quality of life while simultaneously increasing morbidity and mortality. Inspiratory muscle weakness is observed in 30-50% of patients, with the severity of weakness increasing as the disease progresses. Patients exhibit reduced exercise capacity, peripheral and respiratory muscle strength, decreased respiratory function, increased dyspnea, fatigue, and worsened quality of life. However, it is unclear how these parameters will change in patients with inspiratory muscle weakness. Therefore, the study aimed to compare functional exercise capacity, pulmonary function, peripheral muscle strength, dyspnea, fatigue, quality of life and physical activity level in heart failure patients with and without inspiratory muscle weakness and healthy controls

DETAILED DESCRIPTION:
It is believed that respiratory muscle abnormalities develop earlier and more extensively than extremity muscle abnormalities in heart failure. Diaphragm dysfunction contributes to decreased quality of life while simultaneously increasing morbidity and mortality. Inspiratory muscle weakness is observed in 30-50% of patients, with the severity of weakness increasing as the disease progresses. Heart failure patients exhibit increased airway resistance and ventilatory response during exercise. Fatigue and dyspnea are common symptoms associated with exercise intolerance and decreased quality of life in heart failure patients.There is no study in the literature comparing functional exercise capacity, pulmonary function, peripheral muscle strength, dyspnea, fatigue, quality of life and physical activity level in heart failure patients with and without inspiratory muscle weakness (IMW). The aim of the study was to compare functional exercise capacity, pulmonary function, peripheral muscle strength, dyspnea, fatigue, quality of life and physical activity level in heart failure patients with and without IMW and healthy controls.

The study was planned as a cross-sectional, retrospective. Heart failure patient were divided into IMW group or not IMW group due to their MIP values. Also healthy controls who were matched for age-gender were included.

ELIGIBILITY:
Inclusion Criteria:

* HF patients were being aged over18 years
* clinically stable at least four weeks
* having no change in medications over three months

The inclusion criteria for healthy controls were being aged over 18 without a chronic disease

Exclusion Criteria:

* having unstable angina, acute myocardial infarction, uncontrolled hypertension, significant valvular disease, history of malignancy or orthopedic, rheumatologic, neurological, or pulmonary diseases

The exclusion criteria for the healthy controls were having any chronic or systemic disease, and having physical limitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty-one heart failure patients with inspiratory muscle weakness, 30 heart failure patients without inspiratory muscle weakness and 41 healthy controls were included.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | First day
  According to the American Thoracic Society (ATS) guidelines, the 6-minute walk test (6MWT) was used to evaluate functional exercise capacity

SECONDARY OUTCOMES:
Pulmonary function FEV1 | First day
  Pulmonary function FEV1 was assessed by a spirometer according to the ATS/ERS criteria
Pulmonary function FVC | First day
  Pulmonary function FVC was assessed by a spirometer according to the ATS/ERS criteria
Pulmonary function FEV1/FVC | First day
  Pulmonary function FEV1/FVC was assessed by a spirometer according to the ATS/ERS criteria
Pulmonary function PEF | First day
  Pulmonary function PEF was assessed by a spirometer according to the ATS/ERS criteria
Pulmonary function FEF25-75 | First day
  Pulmonary function FEF25-75 was assessed by a spirometer according to the ATS/ERS criteria
Respiratory muscle strength | First day
  Respiratory muscle strength (maximal inspiratory pressure , maximal expiratory pressure; MIP, MEP) was evaluated with a mouth pressure device according to ATS/ERS guidelines.
Peripheral muscle strength | First day
  Peripheral muscle strength was assessed by using a hand-held dynamometer
Dyspnea | First day
  The dyspnea was assessed with The Modified Medical Research Council (MMRC)dyspnea scale. Levels of dyspnea were graded 0-4. Higher scores mean a worse dyspnea level.
Fatigue | First day
  The Fatigue Severity Scale (FSS) was used to identify fatigue. The total score ranges from 0 to 63. Scores above 36 indicate severe fatigue.
The quality of life | Fist day
  Quality of life was evaluated with The Short Form 36 (SF-36) questionnaire. The scores range from 0 to 100. Higher values are indicative of better health.
Physical activity level | First day
  The International Physical Activity Questionnaire (IPAQ) was used to evaluate physical activity level. The total scores of <600 MET-min/week, 600-3000 MET-min/week, and >3000 MET-min/ week were classified as inactive, minimally active, and sufficiently active, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak Güçlü, Prof. Dr, Study Director — Gazi University; Nihan Katayıfçı, Dr., Study Chair — Mustafa Kemal University
Locations (1):
- Gazi University Facutly of Health Sciences Department of Physiotheraphy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lista-Paz A, Langer D, Barral-Fernandez M, Quintela-Del-Rio A, Gimeno-Santos E, Arbillaga-Etxarri A, Torres-Castro R, Vilaro Casamitjana J, Varas de la Fuente AB, Serrano Veguillas C, Bravo Cortes P, Martin Cortijo C, Garcia Delgado E, Herrero-Cortina B, Valera JL, Fregonezi GAF, Gonzalez Montanez C, Martin-Valero R, Francin-Gallego M, Sanesteban Hermida Y, Gimenez Moolhuyzen E, Alvarez Rivas J, Rios-Cortes AT, Souto-Camba S, Gonzalez-Doniz L. Maximal Respiratory Pressure Reference Equations in Healthy Adults and Cut-off Points for Defining Respiratory Muscle Weakness. Arch Bronconeumol. 2023 Dec;59(12):813-820. doi: 10.1016/j.arbres.2023.08.016. Epub 2023 Sep 29. English, Spanish. PMID 37839949
- [Background] Silva Andrade NS, Almeida L, Noronha I, Lima JM, Eriko Tenorio de Franca E, Pedrosa R, Siqueira F, Onofre T. Analysis of respiratory muscle strength and its relationship with functional capacity between different field tests in patients with heart failure. Physiother Theory Pract. 2023 Nov 2;39(11):2427-2437. doi: 10.1080/09593985.2022.2077270. Epub 2022 May 26. PMID 35619283
- [Background] Kasahara Y, Izawa KP, Watanabe S, Osada N, Omiya K. The Relation of Respiratory Muscle Strength to Disease Severity and Abnormal Ventilation During Exercise in Chronic Heart Failure Patients. Res Cardiovasc Med. 2015 Sep 15;4(4):e28944. doi: 10.5812/cardiovascmed.28944. eCollection 2015 Nov. PMID 26528451
- [Background] Miyagi M, Kinugasa Y, Sota T, Yamada K, Ishisugi T, Hirai M, Yanagihara K, Haruki N, Matsubara K, Kato M, Yamamoto K. Diaphragm Muscle Dysfunction in Patients With Heart Failure. J Card Fail. 2018 Apr;24(4):209-216. doi: 10.1016/j.cardfail.2017.12.004. Epub 2017 Dec 28. PMID 29289723
- [Background] Bosnak Guclu M, Bargi G, Katayifci N, Sen F. Comparison of functional and maximal exercise capacity, respiratory and peripheral muscle strength, dyspnea, and fatigue in patients with heart failure with pacemakers and healthy controls: a cross-sectional study. Physiother Theory Pract. 2021 Feb;37(2):295-306. doi: 10.1080/09593985.2019.1630878. Epub 2019 Jun 17. PMID 31204872
- [Derived] Katayifci N, Bosnak Guclu M. Inspiratory muscle weakness further impairs exercise capacity and respiratory functions and increases dyspnea perception in patients with heart failure. Sci Rep. 2025 Sep 1;15(1):32229. doi: 10.1038/s41598-025-16492-6. PMID 40890240